CLINICAL TRIAL: NCT05331118
Title: Perioperative Longitudinal Study of Complications and Long-term Outcomes
Acronym: PLUTO
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, O.L. (Olaf) Cremer, Professor, UMC Utrecht
Other Study IDs: TCBio_19-514
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Perioperative Complication; Infections; Myocardium; Injury; Kidney Injury; Delirium
MeSH Terms: conditions — Infections; Wounds and Injuries; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — EDTA plasma Citrate plasma Serum
  Faeces Oral swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: with an increased risk of complications. Improved preoperative risk stratification and earlier diagnosis of these complications may ameliorate postoperative recovery and improve long-term outcomes. The perioperative longitudinal study of complications and long-term outcomes (PLUTO) aims to establish a comprehensive biorepository that will facilitate research in this field.

Patients undergoing elective intermediate to high-risk non-cardiac surgery are eligible for enrolment. For the first 7 postoperative days (or longer as indicated), participants will be subjected to daily bedside visits by dedicated observers, who adjudicate clinical events and perform non-invasive physiological measurements (including handheld spirometry and single-channel EEG). In addition, we will collect blood samples as well as microbiome specimens at selected time points. Primary study outcomes are the postoperative occurrence of nosocomial infections, major adverse cardiac events, pulmonary complications, acute kidney injury and delirium. Secondary outcomes include mortality as well as long-term psychopathology, cognitive dysfunction, and quality of life.

PLUTO is the first perioperative biobank worldwide that includes a broad range of high-risk surgical patients, collecting prospective bedside data as well as both blood and microbiome specimens during the entire perioperative period. The data and materials collected in PLUTO will be used to develop, externally validate, and update prognostic prediction models for improved risk assessment, to test novel biomarkers for early detection of postoperative complications and to study the aetiology, attributable morbidity and mortality related to these events.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing an elective, high-risk gastro-intestinal or vascular procedure, or intermediate risk procedure (including gynaecological, orthopaedic and head and neck surgery) if the procedure includes a laparotomy and/or is associated with a scheduled hospital length of stay ≥ 5 days.

Exclusion Criteria:

* < 18 years of age
* Emergency surgery
* Severe anaemia (Hb < 4.5 mmol/L)
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing high risk surgery and a selection of intermediate risk procedure as defined by the Surgical Mortality Probability Model. Patients are selected based on procedural risk alone, as we explicitly aim to enrol subjects across a wide range of patient-specific risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2040-02-21 (Estimated); Study Completion 2040-02-21 (Estimated)

PRIMARY OUTCOMES:
Perioperative infectious complications | During hospital admission
  Infectious complications are defined according to Centers for Disease Control and prevention (CDC) criteria and International Sepsis Forum consensus definitions. A comprehensive list of diagnostic criteria, as well as an assessment of the interobserver agreement associated with these, has previously been published in Klein Klouwenberg, Crit Care Med 2013; 41:2373-8. Since these definitions are in agreement with the CDC criteria used in the EPCO definitions, they did not have to be modified for the PLUTO project. For all events, the post hoc probability of true infection will be categorized using a four-point scale (none, possible, probable, and definite infection). This enables us to distinguish cases with true infection from cases with, for example, postoperative systemic inflammation.
Postoperative Pulmonary Complications (PPC) | During hospital admission
  Postoperative pulmonary complications are registered according to the European Perioperative Clinical Outcome (EPCO) definitions. A postoperative pulmonary complication is registered if (1) the patient has a saturation below 90%, (2) the patients oxygen consumption is exceeding 5L/min or (3) the patient's saturation is below 94% while on oxygen therapy. In addition to clinical signs and symptoms, radiology findings, diagnoses and instituted therapies part of the EPCO definitions, duration of the episode and diagnostic modalities used to obtain the diagnosis (e.g. chest x-ray, CT, arterial blood gas, etc.) are registered.
Major Adverse Cardiac Events (MACE) | During hospital admission
  Major Adverse Cardiac Events (MACE) are registered according to the StEP definitions. In addition, the items of the EPCO definition for MACE are included in the registration and all cardiovascular complications included in both these consensus definitions can therefore be reconstructed from the PLUTO database and easily be compared to other perioperative outcome studies. For every patient of 60 years and older, daily troponins are obtained every morning on the first three postoperative days. Daily, an anaesthesiologists assess the troponin values and institutes further diagnostic testing as indicated. For the remaining postoperative days and for patients younger than 60 years of age, troponin is measured on clinical indication.
Acute Kidney Injury (AKI) | During hospital admission
  Acute Kidney Injury (AKI) is defined according to the Risk, Injury, Failure, Loss of kidney function and End-stage kidney disease (RIFLE) criteria. The chart of the patients is assessed on a daily basis for information on urine production and creatinine / kidney function.
Delirium | During hospital admission
  Delirium, defined as either a positive CAM(-ICU) or ≥ 4 points on the AT4.

SECONDARY OUTCOMES:
Complication severity grade | During hosptial admission
  Severity of all surgical complications is assessed according to the Clavien-Dindo classification.
Acute pain | During first 7 days
  Daily pain scores, both in rest and during activity, are measured via the Numeric Rating Scale (NRS). This score ranges from 0 to 10, with 0 being absolutely no pain at all and 10 being the worst imaginable pain.
Long-term psychopathology | At 1 year follow-up
  Long-term psychopathology, defined as symptoms for depression, anxiety and/or post-traumatic stress syndrome (PTSS). Depression is defined as a score ≥ 8 on the HADS-D and anxiety as a score ≥ 8 on the HADS-A. For the IES-R, an item mean score threshold of 1.6 will be used.
Cognitive dysfunction | At 1-year follow-up
  Cognitive dysfunction, as measured by the Cognitive Failure Questionnaire.
Mortality | During first year
  In-hospital mortality, 30-day mortality, one-year mortality and days alive outside of the hospital in the first 30 days following surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: <1 year for the duration of the study

REFERENCES:
- [Derived] de Mul N, Verlaan D, Ruurda JP, van Grevenstein WMU, Hagendoorn J, de Borst GJ, Vriens MR, de Bree R, Zweemer RP, Vogely C, Haitsma Mulier JLG, Vernooij LM, Reitsma JB, de Zoete MR, Top J, Kluijtmans JAJ, Hoefer IE, Noordzij P, Rettig T, Marsman M, de Smet AMGA, Derde L, van Waes J, Rijsdijk M, Schellekens WJM, Bonten MJM, Slooter AJC, Cremer OL. Cohort profile of PLUTO: a perioperative biobank focusing on prediction and early diagnosis of postoperative complications. BMJ Open. 2023 Apr 19;13(4):e068970. doi: 10.1136/bmjopen-2022-068970. PMID 37076142